CLINICAL TRIAL: NCT05688683
Title: Brain Representation of Acquisition in Humans of Motor-Sensory Skills
Acronym: BRAHMS
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: PBN_2022_9
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Epilepsy; Cerebral Tumor
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: use of a theremin-type musical instrument — The patient will perform the task of reproducing sounds by manipulating an object. The settings of the object will be changed and the patient will have to reproduce the sounds a second time by manipulating the object.

SUMMARY:
Interactions between the perceptual and motor systems are fundamental to the performance of complex motor tasks and are at the heart of the fine motor control required for the production of complex sounds such as speech production or playing a musical instrument. In such situations, the brain must learn to generate relevant motor commands to a sound-producing system with fixed physical characteristics, such as the vocal tract or a musical instrument.

No study has yet been able to directly test the dynamic aspect of this sensorimotor learning in an acoustic production task with fine motor control.

The Adolphe de Rothschild Foundation Hospital takes care of patients requiring awake surgery. During these procedures, a direct cortical recording, called electro-corticography, is performed in order to better delineate the tumor or epileptogenic resection area. Reference recordings are made in healthy areas at a distance from the lesion site making it possible to record normal brain activity.

In this case, we would propose to the patient to use a tool similar to the theremin (a musical instrument the size of a golf ball whose displacement in space modulates the frequency and the harmonics of a sound). The patient should therefore learn in order to create relevant motor patterns.

ELIGIBILITY:
Inclusion Criteria:

* Benefiting from an intracranial brain recording during a programmed surgery in awake condition.

Exclusion Criteria:

* Patient with complete deafness
* Patient with a disorder or impairment that does not allow him/her to perform the experimental task according to the investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient benefiting from an intracranial brain recording during a programmed surgery for epilepsy or cerebral tumor resection in awake condition.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
intracranial electroencephalography recording | Day 0
  intracranial electroencephalography recording

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Adolphe de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No